CLINICAL TRIAL: NCT05503901
Title: An Open-Label, Long-Term Phase III Study of STN1012600 Ophthalmic Solution Alone and in Combination With Timolol Ophthalmic Solution, in Subjects With Open Angle Glaucoma or Ocular Hypertension (Angel-J2 Study)
Brief Title: A Long Term Study of STN1012600 in Subjects With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101260006LT
Record Dates: First submitted 2022-08-09; First posted 2022-08-17 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Open Angle Glaucoma, Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: STN1012600 0.002% (Experimental)
  Interventions: Drug: STN1012600 ophthalmic solution 0.002%
- Group 2: STN1012600 0.002% (Experimental)
  Interventions: Drug: STN1012600 ophthalmic solution 0.002%
- Group 3: STN1012600 0.002% + Timolol 0.5% (Experimental)
  Interventions: Drug: STN1012600 ophthalmic solution 0.002% and Timolol ophthalmic solution 0.5%

INTERVENTIONS:
Drug: STN1012600 ophthalmic solution 0.002% — 1 drop STN1012600 ophthalmic solution 0.002% once daily for 52 weeks
  Arms: Group 1: STN1012600 0.002%
Drug: STN1012600 ophthalmic solution 0.002% — 1 drop STN1012600 ophthalmic solution 0.002% once daily for 52 weeks
  Arms: Group 2: STN1012600 0.002%
Drug: STN1012600 ophthalmic solution 0.002% and Timolol ophthalmic solution 0.5% — 1 drop STN1012600 ophthalmic solution 0.002% once daily for 52 weeks and 1 drop Timolol ophthalmic solution 0.5% twice daily for 52 weeks
  Arms: Group 3: STN1012600 0.002% + Timolol 0.5%

SUMMARY:
To evaluate safety and the ocular hypotensive effect of STN1012600 ophthalmic solution 0.002% alone or in combination with Timolol ophthalmic solution 0.5% for 52 weeks in subjects with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of OAG or OHT in both eyes, or one eye with OAG and the other with OHT.
* Corrected Visual Acuity of +0.60 logMAR (Decimal visual acuity 0.3) or better in each eye.

Exclusion Criteria:

* Presence of any active severe external ocular disease, inflammation, or infection of the eye and/or eyelids in either eye.
* History of severe ocular trauma in either eye.
* Any condition that prevents clear visualization of the fundus in either eye.
* Known allergy, hypersensitivity or contraindications to any components of the study medications or other study related procedures/medications.
* History of ocular surgery specifically intended to lower IOP in either eye.
* History of keratorefractive surgery in either eye.
* Females who are pregnant, nursing, or planning a pregnancy.
* Subjects with known or suspected drug or alcohol abuse.
* Participation in other investigational drugs or device clinical trials within 30 days prior to Screening.
* Any decision by the Investigator to terminate a subject in screening or declare any subject ineligible for any sound medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean diurnal intraocular pressure | 52 weeks
  Change from baseline in mean diurnal intraocular pressure at each post-baseline visit
Percent change from baseline in mean diurnal intraocular pressure | 52 weeks
  Percent change from baseline in mean diurnal intraocular pressure at each post-baseline visit

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Kitanagoya Eye Clinic, Aichi
  - Miyake Eye Hospital, Aichi
  - Nagasaka Eye Clinic, Aichi
  - Eto Eye Clinic, Fukuoka
  - Minamoto Eye Clinic, Hiroshima
  - Matsumoto Eye Clinic, Ibaraki
  - IGO Ophthalmic Clinic, Kagoshima
  - Ohguchi Ophthalmic Clinic, Kanagawa
  - Smile Eye Clinic, Kanagawa
  - Inamoto Eye Clinic, Osaka
  - Kubota Eye Clinic, Osaka
  - Nishi Eye Hospital, Osaka
  - Onoe Eye Clinic, Osaka
  - Red Cross Ogawa Hospital, Saitama
  - Nakajima Eye Clinic, Shizuoka
  - Hashida Eye Clinic, Tokyo
  - Seijo Clinic, Tokyo
  - Sinzyuku Eye Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No